CLINICAL TRIAL: NCT04744376
Title: Predictive Value of Quality of Recovery - 15 Questionnaire for Morbidity in Major Abdominal Surgery
Brief Title: Predictive Value of QoR15 for Complications
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mehmet Ali Koç (Other)
Responsible Party: Sponsor-Investigator, Mehmet Ali Koç, MD, Ankara University
Organization: Ankara University (Other)
Other Study IDs: U1111-1264-3497
Record Dates: First submitted 2021-01-29; First posted 2021-02-09 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Complication,Postoperative; Postoperative Period
Keywords: Postoperative morbidity; Postoperaitve mortality; QoR15; ACS risk calculator; Recovery
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Major GIS Surgery: The cohort includes all the patients who undergone major gastrointestinal (GIS) surgery.
  Major GIS surgery includes:
  1. Gastric surgery
  2. Duodenal surgery
  3. Pancreatic surgery
  4. Hepatobiliary surgery
  5. Colonic surgery
  6. Rectal surgery
  Interventions: Other: QoR15; Other: ACS risk calculator; Other: Clavien - Dindo classification

INTERVENTIONS:
Other: QoR15 — Quality of Recovery 15 questionnaire (QoR-15) is a measurement tool that evaluates the recovery quality of patients after surgery and anesthesia by the patient himself.
Other: ACS risk calculator — American College of Surgeons risk calculator is a risk prediction tool for abdominal surgery. It calculates the risk of possible postoperative complications according to the type of surgery, ASA score, and patients' preoperative co-morbidities.
Other: Clavien - Dindo classification — It is a classification for postoperative complications.

SUMMARY:
Surgical operations and recovery after anesthesia is a complex process. Studies examining the interventions performed in the preoperative period often focus on classical clinical outcomes such as postoperative organ dysfunction, morbidity or complications. Postoperative recovery of the patient is rarely considered the most important outcome variable in interventional studies.

In this study, the Quality of recovery 15 (QoR - 15) questionnaire that measures the recovery score, and the American college of surgeons surgical risk calculator have been used to compare the predictive values of patient's preoperative condition on postoperative recovery period and possible morbidity and mortality.

DETAILED DESCRIPTION:
Surgical operations and recovery after anesthesia is a complex process. Studies examining the interventions performed in the preoperative period often focus on classical clinical outcomes such as postoperative organ dysfunction, morbidity or complications. Postoperative recovery of the patient is rarely considered the most important outcome variable in interventional studies. In this study, the effects of both preoperative patient condition and postoperative recovery on morbidity and mortality are investigated.

In order to evaluate the ability of QoR - 15 to predict postoperative complications patients who underwent major abdominal surgery, patients answer the Quality of Recovery 15 questionnaire both in the preoperative and postoperative periods.

In addition, the risk of postoperative complications is calculated in the preoperative period with the American college of surgeons (ACS) surgical risk calculator.

Finally, postoperative complications of all patients are recorded according to Clavien Dindo classification.

The primary goal is to understand the predictive value of the QOR15 score on postoperative complications. Secondarily, it is to compare of predictive values of QoR15 with ACS risk calculator on morbidity and mortality. Another secondary aim is to investigate the effect of preoperative conditions of patients on postoperative recovery.

ELIGIBILITY:
Inclusion Criteria:

All the patients who undergone major GIS surgery

Exclusion Criteria:

1. Patients who has an expected mortality in six months because of the primary disease
2. Patients who received parenteral nutrition before surgery
3. Patients who has a previous major abdominal surgery
4. Patients who do not accept the surgery
5. Patients with a disability who require a nursing care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients who undergone major GIS surgery over age of 18
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Predictive value of QoR - 15 on postoperative complications | In the preoperative period
  QoR - 15 questionnaire is a measurement tool that evaluates the recovery quality of patients after surgery and anesthesia by the patient himself (patient reported outcome measure - PROM). However it has a potential to predict postoperative complication risk.
  Preoperative and postoperative scores of QoR - 15 will be evaluated for a cut-off value regarding postoperative complications which is recorded according to Clavien Dindo classification.
Predictive value of QoR - 15 on postoperative complications | postoperative day 1
  QoR - 15 questionnaire is a measurement tool that evaluates the recovery quality of patients after surgery and anesthesia by the patient himself (patient reported outcome measure - PROM). However it has a potential to predict postoperative complication risk.
  Preoperative and postoperative scores of QoR - 15 will be evaluated for a cut-off value regarding postoperative complications which is recorded according to Clavien Dindo classification.
Predictive value of QoR - 15 on postoperative complications | postoperative day 7
  QoR - 15 questionnaire is a measurement tool that evaluates the recovery quality of patients after surgery and anesthesia by the patient himself (patient reported outcome measure - PROM). However it has a potential to predict postoperative complication risk.
  Preoperative and postoperative scores of QoR - 15 will be evaluated for a cut-off value regarding postoperative complications which is recorded according to Clavien Dindo classification.
Predictive value of QoR - 15 on postoperative complications | postoperative day 30
  QoR - 15 questionnaire is a measurement tool that evaluates the recovery quality of patients after surgery and anesthesia by the patient himself (patient reported outcome measure - PROM). However it has a potential to predict postoperative complication risk.
  Preoperative and postoperative scores of QoR - 15 will be evaluated for a cut-off value regarding postoperative complications which is recorded according to Clavien Dindo classification.

SECONDARY OUTCOMES:
Reliability of QoR - 15 on postoperative complications | In the preoperative period
  QoR15 scores are recorded and the relation of the scores and postoperative complications will be evaluated. After that predictive value of QoR - 15 will be compared to the predictive value of the widely used ACS surgical risk calculator to determine the reliability of QoR - 15 for postoperative complications.
Quality of Recovery | In the preoperative period
  The aim is to investigate the effect of preoperative conditions of patients on postoperative recovery with QoR - 15 questionnaire.
Quality of Recovery | postoperative day 1
  The aim is to investigate the effect of preoperative conditions of patients on postoperative recovery with QoR - 15 questionnaire.
Quality of Recovery | postoperative day 7
  The aim is to investigate the effect of preoperative conditions of patients on postoperative recovery with QoR - 15 questionnaire.
Quality of Recovery | postoperative day 30
  The aim is to investigate the effect of preoperative conditions of patients on postoperative recovery with QoR - 15 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet A Kuzu, MD, Study Director — Ankara University School of Medicine Department of General Surgery; Mehmet A Koç, MD, Principal Investigator — Ankara University School of Medicine Departmernt of General Surgery
Locations (8):
- Turkey (Türkiye) (8):
  - Çukurova University School of Medicine Department of General Surgery, Adana
  - Ankara University School of Medicine Department of General Surgery, Ankara
  - Diskapi Research and Training Hospital, Ankara
  - Hacettepe University School of Medicine Department of General Surgery, Ankara
  - Ministry of Health Ankara City Hospital, Ankara
  - Antalya Research and Trainig Hospital, Antalya
  - Ataturk University School of Medicine Department of General Surgery, Erzurum
  - Ministry of Health Kayseri City Hospital, Kayseri

IPD SHARING:
Plan to Share IPD: No